CLINICAL TRIAL: NCT03730103
Title: Evaluating Safety, Cost, and Patient Satisfaction With Same Day Discharge After Minimally-invasive Sacrocolpopexy
Brief Title: Same Day Discharge After Minimally-invasive Sacrocolpopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-563
Record Dates: First submitted 2018-10-21; First posted 2018-11-05 (Actual); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-06

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: Prospective cohort study with historical controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Historical control group (No Intervention): The investigators will use data from a historical control group discharged on POD 1 after minimally invasive sacrocolpopexy to examine Aim 1 and Aim 2. This is a cohort of 60 women matching our eligibility criteria from a prospective randomized trial of two different types of lightweight polypropylene mesh (IRB #14-354). This study completed recruitment 2017. It consists of a group of women who underwent minimally invasive sacrocolpopexy using the same surgical approaches, at the same institutions
- Same day discharge group (Experimental): 47 women will be recruited for same day discharge after laparoscopic sacrocolpopexy. We will compare aim 1 and 2 (serious adverse events and procedure-related costs) between the two groups
  Interventions: Other: Same day discharge

INTERVENTIONS:
Other: Same day discharge — Patients will be discharged home from the hospital on the day of her surgery.
  Arms: Same day discharge group

SUMMARY:
This is a prospective cohort study evaluating safety, cost and patient satisfaction with SDD for patients undergoing minimally invasive sacrocolpopexy for pelvic organ prolapse. A prospectively collected, historical control group who underwent the same surgical procedure will be utilized to compare these outcomes when applicable. SDD will be facilitated in part by a utilizing novel patient education video created for this study and implementing an ERAS pathway. All patients meeting eligibility criteria will be approached for study participation. Outcomes will be assessed on POD 0/1 and at the routine post-operative follow up visit, generally at 6 weeks after surgery.

DETAILED DESCRIPTION:
Enhanced recovery after surgery (ERAS) pathways play a critical role in the delivery of high-quality surgical care. These protocols incorporate multiple perioperative patient interventions including preemptive analgesia, measures to reduce postoperative nausea and emesis, fluid balance aimed at euvolemia, and both early ambulation and oral intake. ERAS pathways are significant because they have been shown to shorten recovery, decrease hospital stay, reduce complications/nosocomial infections, and conserve resources.1-20 Same-day discharge (SDD) is a central aspect of enhanced recovery pathways.

SDD and ERAS protocols are part of a new initiative within the Women's Health Institute, and their application for gynecologic surgery is of increasing interest across the country.1-19 To date, the focus of studies has largely been on laparoscopic and robotic hysterectomy in the benign and gynecologic oncology literature. Studies have consistently demonstrated both feasibility and safety of SDD after laparoscopic and robotic hysterectomy, with no significant increase in complications or readmissions as compared to discharge on postoperative day (POD) 1. In fact, a recent systematic review by Korsholm et al of 15 observational studies with nearly 12,000 patients revealed SDD is feasible, at a rate of nearly 80%, when patients are properly selected and careful surgical planning is performed.3 Studies have also demonstrated high patient satisfaction10,12 and less cost18 with SDD after minimally invasive hysterectomy. SDD has been applied in other minimally invasive gynecologic procedures, such as minimally invasive myomectomy, with low readmission rates (0.6% within 48 hours, 1.4% over 3 months).20

ERAS pathways can have an important role in other areas of gynecologic surgery. In the field of urogynecology, quality of life reconstructive surgery is often performed to address symptoms of pelvic organ prolapse, urinary incontinence, and/or fecal incontinence. A prospective study by Kalogera et al evaluated the impact of an ERAS pathway for patients undergoing vaginal reconstructive surgeries for pelvic organ prolapse versus historical controls.21 In this cohort, patient satisfaction with perioperative care was high, mean duration of hospital stay was significantly reduced, and there were no differences in 30 day outcomes. In a case series by Zakaria and Levy, an ERAS pathway was utilized after vaginal hysterectomy, which permitted SDD in 96% of patients.19 Notably, only 5 of the 1071 patients required readmission or emergency room evaluation within 30 days of surgery. Taken together, these studies provide support for the application of ERAS pathways in urogynecology, where well-selected surgical candidates are undergoing surgeries appropriate for SDD.

Yet, to date, only one research study has investigated the role of SDD after minimally invasive sacrocolpopexy. A sacrocolpopexy is a surgery for pelvic organ prolapse in which a bridging piece of mesh is utilized to suspend the vaginal cuff to the anterior longitudinal ligament overlying the sacral promontory. This is an extensively studied and highly effective surgical technique to correct pelvic organ prolapse and is a mainstay in the field of urogynecology. A study by Faucheron et al evaluated SDD for robotic and laparoscopic ventral rectopexy, a similar mesh-augmented procedure that is performed for rectal prolapse, and concluded that SDD is feasible and safe.22 A preliminary study by Lloyd et al performed at the Cleveland Clinic within the Female Urology division investigated SDD after minimally invasive sacrocolpopexy (article in press). In this study, SDD was achieved in 10 of 12 patients (83.3%). The two patients who did not have SDD were due to case completion after 6PM, a preset case completion requirement. Outcomes were also retrospectively compared between patients who underwent SDD (N= 10) and patients who stayed overnight (N=30). Only one patient had an emergency department visit on POD 20, due to an unrelated mechanical fall. Importantly, there were no major complications in either group requiring procedural interventions, new prescriptions, or additional interventions. Recently, a study by Kisby et al was published examining SDD after robotic-assisted sacrocolpopexy. In this retrospective study, 80 women underwent SDD compared to 192 who were discharged on >/=POD 1.23 This study found no difference in unplanned provider visits, emergency department visits or readmissions between the groups.

The investigators hypothesize that an ERAS protocol utilizing SDD for minimally invasive sacrocolpopexy is as safe as those that utilize discharge on POD 1 while incurring less total procedure-related costs and being acceptable as a post-op management plan for patients. The objective of this study is to provide data which are necessary to widely implement SDD after a minimally invasive sacrocolpopexy. The results of this research will have a significant impact on increasing patient satisfaction, minimizing resource utilization, and improving clinical practice patterns in the field of urogynecology, both for this procedure and potentially other surgeries within our subspecialty.

Specific Aims Aim 1. To compare the incidence of adverse events in patients following a SDD protocol for minimally invasive sacrocolpopexy compared to those patients discharged on POD 1.

The investigators hypothesize that there is no difference in the incidence of adverse events between SDD compared to discharge on POD 1 after minimally invasive sacrocolpopexy. Using the Epic electronic medical record (EMR), the investigators will evaluate 1) the number of unscheduled office visits, patient-initiated calls for a surgery-related complication, emergency department visits, and readmissions/reoperations of patients who had a SDD protocol and 2) the severity of any adverse events using the Clavien Dindo Scale. The investigators will utilize patient phone calls to inquire about any of the aforementioned events outside of our institution. The investigators will compare incidence of postoperative adverse events between patients undergoing SDD versus a historical control group who were discharged on POD 1.

Aim 2. To compare the total procedure-related costs associated with SDD compared to discharge on POD 1 for minimally invasive sacrocolpopexy.

The investigators hypothesize that the total costs associated with SDD following minimally invasive sacrocolpopexy is less than the same procedure with discharge on POD 1. The investigators will utilize data from the billing function of Epic EMR to compare total procedure-related costs for each approach to minimally invasive sacrocolpopexy.

Aim 3. To determine patient satisfaction with SDD after minimally invasive sacrocolpopexy.

The investigators hypothesize that patients will be satisfied with SDD after minimally invasive sacrocolpopexy. The investigators plan to address this aim using a series of validated measures.

ELIGIBILITY:
Inclusion Criteria:

* Age <80 years old
* Preoperative American Society of Anesthesiologists grade I (normal healthy patient) or II (mild systemic disease)
* Access to ancillary care, including phone advice, nurse and outpatient clinic numbers
* Caretaker at home for at least 24 hours post-operatively
* Able to speak and read English
* Has decision-making capacity and able to provide consent for research participation

Exclusion Criteria:

* Laparoscopic, robotic, or open abdominal surgical procedures that require an overnight admission. This may be due to unanticipated additional intraoperative procedures or surgical complications such as unintentional cystotomy or enterotomy, hemorrhage, or anesthetic complication.
* Patients undergoing concomitant laparoscopic colorectal procedures or anal sphincteroplasty
* Surgery start time after 1:00PM, as previous studies have determined this is associated with a decreased likelihood of SDD3,14
* Pregnancy or positive hCG testing, which is standard of care preoperative testing

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All participants are women having surgery for pelvic organ prolapse
Enrollment: 52 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa C Hickman, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be made available to other researchers

REFERENCES:
- [Derived] Hickman LC, Paraiso MFR, Goldman HB, Propst K, Ferrando CA. Same-Day Discharge After Minimally Invasive Sacrocolpopexy Is Feasible, Safe, and Associated With High Patient Satisfaction. Female Pelvic Med Reconstr Surg. 2021 Aug 1;27(8):e614-e619. doi: 10.1097/SPV.0000000000000998. PMID 33411456

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were excluded: (2) case start-times after 1:00 p.m., (1) case aborted, (1) approach changed to vaginal, (1) patient withdrew.
Period: Overall Study
Arm/Group | Historical Control Group | Same Day Discharge Group
Started | 61 | 52
Completed | 61 | 47
Not Completed | 0 | 5
Not completed — Did not meet inclusion criteria | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Historical Control Group | Same Day Discharge Group | Total
Number analyzed (Participants) | 61 | 47 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 29 | 70
  >=65 years | 20 | 18 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (8.0) | 62.2 (8.9) | 61.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 47 | 108
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 58 | 45 | 103
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 61 | 47 | 108

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants* With Serious Adverse Events
Description: The investigators wish to compare the incidence of adverse events in patients following a SDD protocol for minimally invasive sacrocolpopexy compared to those patients discharged on POD 1.
Time Frame: 6 weeks postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Control Group | Same Day Discharge Group
Number analyzed (Participants) | 61 | 47
Participants | 4 | 3

2. Secondary Outcome: Number of Participants With One or More Patient- Initiated Phone Calls
Description: The incidence of patient-initiated phone calls for a surgery-related complication in patients following a SDD protocol for minimally invasive sacrocolpopexy compared to those patients discharged on POD 1.
Time Frame: 6 weeks postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Control Group | Same Day Discharge Group
Number analyzed (Participants) | 61 | 47
Participants
  1 phone call | 16 | 9
  2 phone calls | 20 | 7
  3 phone calls | 7 | 4
  4+ phone calls | 1 | 3

3. Secondary Outcome: Number of Participants With One or More Unscheduled Office Visits, Including Voiding Trials
Description: The incidence of unscheduled office visits, including voiding trials, for patients following a SDD protocol for minimally invasive sacrocolpopexy compared to those patients discharged on POD 1.
Time Frame: 6 weeks postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Control Group | Same Day Discharge Group
Number analyzed (Participants) | 61 | 47
Participants
  1 office visit | 14 | 14
  2 office visits | 3 | 3
  3 office visits | 0 | 3

4. Secondary Outcome: Number of Participants With One or More Emergency Department Visits
Description: The incidence of emergency department visits for patients following a SDD protocol for minimally invasive sacrocolpopexy compared to those patients discharged on POD 1.
Time Frame: 30 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Control Group | Same Day Discharge Group
Number analyzed (Participants) | 61 | 47
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: 6-weeks
Arm/Group | Historical Control Group | Same Day Discharge Group
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/47
Serious Adverse Events (participants affected / at risk) | 4/61 | 3/47
Other Adverse Events (participants affected / at risk) | 0/61 | 0/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Historical Control Group (N=61) | Same Day Discharge Group (N=47)
Wound infection (Infections and infestations) | 1 (1) | 2 (2)
Bowel obstruction (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiopulmonary (Cardiac disorders) | 1 (1) | 0 (0)
Neurologic injury (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT03730103/Prot_SAP_000.pdf